CLINICAL TRIAL: NCT03176498
Title: The Effects of Human Umbilical Cord Mesenchymal Stem Cell Therapy on Neurological Function for Cerebral Infarction Patients in Convalescent Period.
Brief Title: Human Umbilical Cord Mesenchymal Stem Cell Therapy (19#iSCLife®-CI) for Cerebral Infarction Patients in Convalescent Period.
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Others
Sponsor: Sclnow Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCLnow-IMIMH-01
Record Dates: First submitted 2017-05-23; First posted 2017-06-05 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Infarction
Keywords: cerebral Infarction; umbilical cord mesenchymal stem cells
MeSH Terms: conditions — Cerebral Infarction | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Basic medication：Aspirin Enteric-coated Tablets & Atorvastatin Calcium； Allogeneic umbilical cord mesenchymal stem cells
  Interventions: Biological: Allogeneic umbilical cord mesenchymal stem cell; Drug: Aspirin Enteric-coated Tablets & Atorvastatin Calcium
- Control group (Placebo Comparator): Basic medication：Aspirin Enteric-coated Tablets & Atorvastatin Calcium; Placebo：saline
  Interventions: Drug: Aspirin Enteric-coated Tablets & Atorvastatin Calcium

INTERVENTIONS:
Biological: Allogeneic umbilical cord mesenchymal stem cell — Experimental group receive Allogeneic umbilical cord mesenchymal stem cell，i.v (SCLnow 19#)
  Arms: Experimental group
Drug: Aspirin Enteric-coated Tablets & Atorvastatin Calcium — Aspirin Enteric-coated Tablets, 0.1g/d by mouth; Atorvastatin Calcium, 20mg/d by mouth.

SUMMARY:
This is a randomized, double-blind study. Human umbilical cord mesenchymal stem cells (hUC-MSC) will be treated on cerebral infarction patients, and evaluates their neurological function of convalescent period.

DETAILED DESCRIPTION:
40 participants will be selected based on eligibility criteria and collected information, then, randomly separated into two groups. All participants will sign informed consent form, monitor vital signs, laboratory examination (CT/MRI, blood routine examination, urine routine examination, liver function, renal function, etc.), NIHSS, Fugl-Meyer analysis (FMA) 0-3 days before treatment. All of them will receive basic treatment with Aspirin Enteric-coated Tablets and Atorvastatin Calcium. And experimental group will treat with hUC-MSC, control group with placebo (normal saline) on the 7th and 14th day. After the treatment, investigator will follow-up, monitor vital signs, laboratory examination, NIHSS, FMA analysis on 2 weeks, 1 month, and 6 months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* proved cerebral infarction by CT or MRI.
* no cerebrovascular disease before
* signed informed consent form

Exclusion Criteria:

* serious body and intracranial lesions (tumor, infection, etc.)
* patients repeated cerebral infarction attacks
* multi-foci of cerebral infarction
* history of drug dependence and mental disease
* disturbance of consciousness and non-compliance patients
* subjects who are HIV positive
* pregnant or lactation
* donor: HIV infected, Active hepatitis B/C infected, Syphilis antibody positive
* subjects/ donor: alcoholism, drug addicts or mental disease

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Motor function analysis | 6 months
  Based on Activity of Daily Living Scale (ADL) to analysis efficacy of cell treatment.The score of patient with upper limb >60, and total score >90 is considered good recovery.

SECONDARY OUTCOMES:
Neurological deficits analysis | 6 months
  According to Chinese scale of clinical neurologic deficit to analysis, the result as follow:
  * Excellent: after treatment, patient with consciousness, and clinical symptoms improved;
  * Effective: vital signs and main symptoms in remission;
  * Inefficient: no obvious improvement or condition worsened.
Limb motor function analysis | 6 months
  Using fugl-meyer assessment evaluate motor function. Mild movement disorder: 96 - 99; Moderate movement disorder: 85 - 95; Obvious movement disorder: 50 - 84; Serious movement disorder: < 50
Barthel Index analysis | 6 months
  Obvious effective: Barthel Index score between 96 - 99, patient with self care ability.
  Effective:Barthel Index score between 70 - 89, patient with condition improved. Invalid: The effect do not meet above standards.

CONTACTS AND LOCATIONS:
Overall Officials: Wulan, Study Director — Inner Mongolia International Mongolian Hospital; Lei Guo, Dr, Study Chair — China-Japan Union Hospital, Jilin University
Locations (1):
- Inner Mongolia International Mongolian Hospital, Hohhot, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: No